CLINICAL TRIAL: NCT02350712
Title: An Open Label, Phase 1B Safety Evaluation of Patritumab (U31287) in Combination With Cetuximab Plus Platinum Containing Therapy In Subjects With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Patritumab With Cetuximab and a Platinum Containing Therapy for Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U31287-A-U106; 2014-002445-22 (EudraCT Number)
Record Dates: First submitted 2015-01-19; First posted 2015-01-30 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Recurrent or metastatic squamous cell carcinoma of the head and neck; SCCHN
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence | interventions — patritumab; Antibodies, Monoclonal; Cetuximab; Drug Therapy; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- All Participants - Period 1 (Experimental): All participants receive patritumab with cetuximab plus platinum-based therapy (cisplatin or carboplatin) in Period 1 - Initial phase of the trial.
  Interventions: Drug: Patritumab; Drug: Cetuximab; Drug: Cisplatin; Drug: Carboplatin
- All Participants - Period 2 (Experimental): Participants deriving clinical benefit enter Period 2 - Extension phase, during which they continue to receive patritumab with cetuximab, but not platinum-based therapy.
  Interventions: Drug: Patritumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Patritumab — Patritumab initial loading dose is 18 mg/kg IV over 60 minutes, followed in Cycle 2 and beyond with a maintenance dose of 9 mg/kg IV over 60 minutes (+/- 10 minutes) every 3 weeks. Infusion time can be extended to a maximum of 120 minutes for participants unable to tolerate the 60-minute infusion.
  Other Names: U3-1287; Monoclonal antibody
Drug: Cetuximab — Cetuximab initial dose at 400 mg/m2 IV as a 2-hour infusion, followed by 250 mg/m2 IV over 60 minutes weekly.
  Other Names: Chemotherapy
Drug: Cisplatin — Cisplatin is given as an IV infusion, over 1 hour, 1 hour after the cetuximab infusion, every 3 weeks up to a maximum of 6 cycles (with standard pre- or post-treatment therapies at the investigator's discretion).
  Other Names: Chemotherapy; Platinum therapy
  Arms: All Participants - Period 1
Drug: Carboplatin — Carboplatin is given as an IV-bolus, over 30-60 minutes, every 3 weeks, for a maximum of 6 cycles (with standard pre- or post-treatment therapies at the investigator's discretion).
  Other Names: Chemotherapy; Platinum therapy
  Arms: All Participants - Period 1

SUMMARY:
The purpose of this study is to test a study drug called patritumab. Patritumab may work when combined with other medications that are approved in the UK for treating Squamous Cell Carcinoma of the Head and Neck (SCCHN), called cetuximab, cisplatin or carboplatin. It is hoped that patritumab may have some benefit in treating patients with cancer. This study will help identify how much patritumab can be given in combination with cetuximab, and cisplatin or carboplatin. This study will show how safe and how well tolerated patritumab is when these medications are given together.

DETAILED DESCRIPTION:
The trial will be performed in two "phases" (Periods):

Period 1: Initial phase in which the recommended phase 2 dose (RP2D) is determined

Period 2: Extension phase in which participants who are deriving benefit (stable disease or better) will have the opportunity to continue treatment at the discretion of the Investigator

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent disease or metastatic SCCHN originating from the oral cavity, oropharynx, hypopharynx, and larynx
* Has documented disease recurrence following prior treatment
* Has Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Has adequate hematological function, per protocol
* Has adequate renal function, per protocol
* Has adequate hepatic function, per protocol
* Has prothrombin time (PT) or partial thromboplastin time (PTT) within 1.5 x upper limit of normal (ULN)
* Has a negative serum pregnancy test performed within 14 days prior to enrollment (where required by local regulations, test may be required within 72 hours prior to enrollment), if a woman of child-bearing potential
* Agrees to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after last study dose received, if of child-bearing potential
* Is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Has left ventricular ejection fraction (LVEF) < 50%
* Has received prior epidermal growth factor receptor (EGFR) targeted regimen
* Has received prior anti-HER2, anti-HER3, or anti-HER4 therapy
* Has received prior treatment for recurrent/metastatic disease
* Has history of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
* Has known history of and active brain metastases
* Has uncontrolled hypertension (systolic > 160 mm Hg or diastolic > 100 mm Hg)
* Has clinically significant electrocardiogram (ECG) changes
* Has had myocardial infarction within 1 year before enrollment, symptomatic congestive heart failure (New York Heart Association >Class II), unstable angina, or unstable cardiac arrhythmia requiring medication
* Had platinum-containing drug therapy/chemotherapy with radiotherapy < 6 months before study drug treatment
* Had therapeutic or palliative radiation therapy or major surgery within 4 weeks before study drug treatment.
* Participated in clinical drug trials within 4 weeks before study drug treatment or is currently participating in other investigational procedures
* Has uncontrolled infection requiring intravenous (IV) antibiotics, antivirals, or antifungals, known human immunodeficiency virus (HIV) infection, active hepatitis B or C infection, or is undergoing medical treatment for infection
* Has uncontrolled type 1 or 2 diabetes mellitus
* Has known hypersensitivity or allergic reaction against any of the components of the trial treatment
* Is pregnant, breastfeeding, or unwilling/unable to use acceptable contraception
* Has psychological, social, familial, or geographical factors that would interfere with study participation or follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Percentage of participants experiencing dose-limiting toxicities (DLTs) | 6 months
  DLTs are used to determine the maximum tolerated dose.

SECONDARY OUTCOMES:
Pharmacokinetic profile of serum patritumab | 6 months
  Cmax and AUC
Pharmacokinetic profile of serum cetuximab | 6 months
  Cmax and AUC
Percentage of participants with human anti-human antibody (HAHA) formation (anti-patritumab antibodies) | 6 months
Titer of HAHA formation (anti-patritumab antibodies) | 6 months
  A titer is a way of expressing concentration. Titer testing employs serial dilution to obtain approximate quantitative information from an analytical procedure that inherently only evaluates as positive or negative. The titer corresponds to the highest dilution factor that still yields a positive reading.

CONTACTS AND LOCATIONS:
Overall Officials: Global Team Leader, Study Director — Daiichi Sankyo
Locations (3):
- United Kingdom (3):
  - The Royal Marsden Hospital, Sutton, Surrey
  - University College London Hospital, London
  - The Royal Marsden Hospital, London